CLINICAL TRIAL: NCT06142318
Title: Application of Pirfenidone as a Radiosensitizer in the Treatment of Head and Neck Squamous Cell Carcinoma: Phase II Clinical Study
Brief Title: Pirfenidone as a Radiosensitizer in the Treatment of Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NFEC-2023-477
Record Dates: First submitted 2023-11-16; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Radiotherapy; Radiosensitizer; Pirfenidone
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pirfenidone group (Experimental): Calculate from 2 weeks before the start of radiotherapy: week 1: pirfenidone 200mg, tid; week 2: pirfenidone 400mg tid; during radiotherapy: pirfenidone 600mg tid.
  Interventions: Drug: Pirfenidone
- Control group (Placebo Comparator): Calculate from 2 weeks before the start of radiotherapy: week 1: placebo 200mg, tid; week 2: placebo 400mg tid; during radiotherapy: placebo 600mg tid.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pirfenidone — Dose climbing started two weeks before the start of radiotherapy, and the maintenance dose of 600mg bid was reached in the third week until the end of radiotherapy.
  Arms: Pirfenidone group
Drug: Placebo — Dose climbing started two weeks before the start of radiotherapy, and the maintenance dose of 600mg bid was reached in the third week until the end of radiotherapy.
  Arms: Control group

SUMMARY:
Head and neck squamous cell carcinoma (HNSCC) is the sixth most common cancer worldwide, with a 5-year survival rate of less than 50%. Radiotherapy is an important measure to control tumor recurrence. Although radiotherapy has been widely used in patients with head and neck squamous cell carcinoma, the 2-year local recurrence rate of patients with locally advanced disease is still as high as 50%-60%, and the distant metastasis rate is as high as 20%-30%. This is associated with a lower radiosensitivity in HNSCC. Our previous study has confirmed that type I collagen secreted by cancer-associated fibroblasts (CAFs) can enhance the radioresistance of head and neck squamous cell carcinoma. We also confirmed that pirfenidone could reduce type I collagen expression in CAFs and enhance radiosensitivity in vitro and in vivo. Therefore, we plan to translate the basic research into clinical practice and conduct a prospective interventional phase II clinical trial to investigate the safety and efficacy of pirfenidone as a radiosensitizer in HNSCC.

ELIGIBILITY:
Inclusion Criteria:

1. be at least 18 years old;
2. provide written informed consent;
3. head and neck squamous cell carcinoma confirmed by biopsy (2022 WHO criteria);
4. no previous head and neck radiotherapy;
5. The presence of measurable lesions: no surgical treatment or postoperative imaging evaluation indicated that the tumor was not completely resected;
6. ECOG PS: 0/1;
7. Laboratory confirmation of good organ function. It should be given within 10 days before the first dose of treatment; 8) expected survival time ≥3 months.

Exclusion Criteria:

1. no indications for or contraindications to radiotherapy after evaluation;
2. no oral medication;
3. pregnancy or lactation;
4. patients with known allergy to pirfenidone or other contraindications;
5. concurrent tumors (except cured basal cell or squamous cell skin cancer, and cervical cancer in situ);
6. patients had any serious coexisting medical conditions that could pose an unacceptable risk or negatively affect trial adherence. "For example, unstable heart disease requiring treatment, chronic hepatitis, kidney disease, poor condition, uncontrolled diabetes (fasting blood glucose > 1.5 × ULN), and mental illness."

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1 month
  The objective response rate (ORR) is the proportion of patients who achieve a prespecified reduction in tumor volume that is maintained for a minimum duration. The objective response rate was defined as the sum of complete response plus partial response (CR+PR). According to RECIST1.1 criteria, CR was defined as the disappearance of target lesions and the reduction of the short diameter of pathological lymph nodes to less than 10mm. PR: the sum of the measured diameters of the target lesions reduced by 30% compared with the baseline; PD: the sum of the major diameters of all target lesions increased by at least 20%, and the absolute value of the sum of the major diameters increased by more than 5mm, or new lesions appeared. SD: Changes between PR and PD.

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
  OS was defined as the time from the date of inclusion until death from any cause.
Incidence of Treatment-Emergent Adverse Events | During treatment and 12 weeks after treatment
  treatment-related adverse events will be assessed by CTCAE v5.0

OTHER OUTCOMES:
the biomarkers correlated with ORR and OS | 2 years
  The correlations between ORR, OS and cancer associated fibroblasts, collagen type I, PD-L1 expression in tissues, tumor mutation burden, tumor-related gene changes, plasma cytokines or other biomarkers were explored.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Southern medical university, Guangzhou, Guangdong
  - Fujian Provinical Hospital, Fuzhou
  - Huizhou Central People's Hospital, Huizhou
  - Jieyang people's hospital, Jieyang
  - Meizhou People's Hospital, Meizhou Academy of Medical Sciences Meizhou, Meizhou

IPD SHARING:
Plan to Share IPD: No